CLINICAL TRIAL: NCT06658106
Title: Effect of Thera-Band Elastic Band-Assisted Progressive Resistance Training on Physical Health and Frailty Status in Patients with Diabetes Mellitus Complicated by Frailty Syndrome: a Randomized Controlled Trial
Brief Title: Effect of Thera-Band Elastic Band-Assisted Progressive Resistance Training on Physical Health in Diabetes Patients with Frailty Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Rongjun Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023 LSY No. (8)
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Frailty Syndrome; Progressive Resistance Training; Thera-Band Elastic Band
MeSH Terms: conditions — Diabetes Mellitus; Frailty

STUDY DESIGN:
Intervention Model Description: This clinical trial will utilize a parallel study design, wherein participants will be randomly assigned to one of two groups: the research group receiving Thera-Band elastic band-assisted progressive resistance training (PRT) and the control group receiving conventional diabetes management. Each group will be treated independently throughout the study duration of 12 weeks. The outcomes of interest will be assessed at baseline and after the intervention period to determine the effectiveness of the exercise program in improving physical health and reducing frailty in older adults with diabetes mellitus. This design allows for a direct comparison between the intervention and control groups, providing robust data on the efficacy of the Thera-Band PRT approach.
Masking Description: In this clinical trial, there will be no masking of participants, care providers, investigators, or outcomes assessors. All parties involved will be aware of the interventions assigned to participants. This decision was made to facilitate adherence to the Thera-Band elastic band-assisted progressive resistance training program and to ensure that the research team can monitor the participants effectively throughout the intervention. While this approach allows for clear communication and immediate feedback regarding the exercise protocol, it may introduce bias in the assessment of outcomes. However, objective measures such as blood glucose levels and physical performance assessments will be used to minimize this potential bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thera-Band Elastic Band-Assisted Progressive Resistance Training Group (Experimental): In the Thera-Band Elastic Band-Assisted Progressive Resistance Training Group, participants will engage in a structured exercise program utilizing Thera-Band elastic bands for resistance training. The intervention will occur three times a week for 12 weeks, with each session lasting approximately 50 minutes. Exercises will target major muscle groups, including upper and lower limbs, and will be designed to improve strength, balance, and overall physical function. Participants will be instructed to exercise at 60%-80% of their maximum heart rate to ensure an effective training intensity. The program aims to enhance physical health, reduce frailty, and improve quality of life for older adults with diabetes mellitus and frailty syndrome. Participants will receive guidance from trained exercise instructors and will be monitored for any adverse reactions during the training sessions.
  Interventions: Behavioral: Thera-Band Elastic Band-Assisted Progressive Resistance Training; Behavioral: Conventional Diabetes Management
- Conventional Diabetes Management Group (Active Comparator): In the Conventional Diabetes Management Group, participants will receive standard care for diabetes management, which includes basic health education and guidance on diet, exercise, medication adherence, and daily care practices. This group will not engage in the Thera-Band exercise program but will continue their usual activities and follow-up care as prescribed by their healthcare providers. The aim of this arm is to provide a comparison to the experimental group regarding the effectiveness of the elastic band-assisted progressive resistance training on physical health and frailty outcomes. Participants will be monitored for their blood glucose levels and overall health status throughout the study period, and any changes in their condition will be documented.
  Interventions: Behavioral: Conventional Diabetes Management

INTERVENTIONS:
Behavioral: Thera-Band Elastic Band-Assisted Progressive Resistance Training — Thera-Band Elastic Band-Assisted Progressive Resistance Training: This intervention involves a structured exercise program using Thera-Band elastic bands for resistance training, conducted three times a week for 12 weeks. Each session lasts approximately 50 minutes and includes exercises targeting major muscle groups, such as upper arms, shoulders, chest, lumbar, and lower limbs. Participants will perform each exercise for 8-12 repetitions in 2-3 sets with 1-minute intervals, aiming for an intensity of 60%-80% of their maximum heart rate. The program is designed to improve strength, balance, and overall physical function, thereby reducing frailty in older adults with diabetes.
  Arms: Thera-Band Elastic Band-Assisted Progressive Resistance Training Group
Behavioral: Conventional Diabetes Management — Conventional Diabetes Management: Participants in this arm will receive standard care for diabetes management, which includes health education covering diet, medication adherence, exercise recommendations, and routine health monitoring. This arm serves as a comparator to assess the effectiveness of the progressive resistance training intervention.

SUMMARY:
Goal: The goal of this clinical trial is to evaluate the effectiveness of Thera-Band elastic band-assisted progressive resistance training (PRT) in improving physical health and reducing frailty in older adults with diabetes mellitus (DM) complicated by frailty syndrome (FS).

Main Questions:

Does Thera-Band elastic band-assisted PRT lower blood glucose levels in patients with DM? Does Thera-Band elastic band-assisted PRT improve physical function, as measured by handgrip strength and gait speed, in patients with FS? If there is a comparison group: Researchers will compare the Thera-Band elastic band PRT group to the conventional treatment group to see if the PRT intervention leads to greater improvements in physical health and frailty status.

Participants will:

Undergo Thera-Band elastic band-assisted progressive resistance training for 12 weeks, attending sessions three times a week.

Complete assessments of their blood glucose levels and physical function before and after the intervention.

Provide feedback on their fatigue, psychological state, and any adverse reactions during the training period.

DETAILED DESCRIPTION:
This clinical trial aims to assess the effects of Thera-Band elastic band-assisted progressive resistance training (PRT) on the physical health of patients with diabetes mellitus (DM) complicated by frailty syndrome (FS). The trial will involve 96 participants aged 60 years and older, diagnosed with type 2 DM and identified as frail based on the Tilburg Frailty Indicator (TFI).

Participants will be randomly assigned to either the research group, receiving Thera-Band PRT, or a control group receiving conventional diabetes management. The PRT sessions will occur three times a week for 12 weeks, focusing on strength training exercises targeting major muscle groups using elastic bands of varying resistance. Training sessions will include upper and lower body exercises, ensuring participants work at 60%-80% of their maximum heart rate.

Primary outcomes will include changes in fasting blood glucose levels, handgrip strength (HS), and usual gait speed (UGS), assessed before and after the intervention. The Short Physical Performance Battery (SPPB) will evaluate overall physical function, while the FRAIL scale will assess frailty status. Psychological assessments will be conducted using the Geriatric Depression Scale-15 (GDS-15) and the Diabetes Distress Scale (DDS) to measure mental well-being.

Adverse events, such as injuries or discomfort during training, will be monitored throughout the study to ensure participant safety. This trial will contribute valuable clinical evidence regarding the effectiveness of elastic band-assisted PRT in enhancing physical health and reducing frailty in older adults with diabetes, ultimately informing best practices for managing this vulnerable patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus (T2DM).
* Fasting blood glucose level of less than 16.7 mmol/L.
* Frailty score of 4 points or higher on the Tilburg Frailty Indicator (TFI).
* Aged 60 years or older.
* Muscle strength rated at level 4 or higher.
* No participation in regular exercise in the past.

Exclusion Criteria:

* Presence of serious heart conditions, such as severe heart failure or significant heart disease.
* Loss of consciousness (e.g., being excessively sleepy or in a coma).
* Diagnosis of severe Alzheimer's disease or other significant cognitive impairments.
* Physical disabilities that would prevent participation in exercise.
* Diagnosis of severe osteoporosis (weak bones).
* Communication barriers that prevent understanding or cooperation with the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Handgrip Strength | From enrollment to the end of treatment at 12 weeks.
  Measured using an electronic hand muscle developer to assess muscle strength and physical function at baseline and after the 12-week intervention period.
Usual Gait Speed | From enrollment to the end of treatment at 12 weeks.
  Assessed using the 6-minute walk test to evaluate mobility and physical performance before and after the intervention.

SECONDARY OUTCOMES:
Short Physical Performance Battery | From enrollment to the end of treatment at 12 weeks.
  Evaluated at baseline and after 12 weeks to measure balance, walking ability, and sit-to-stand performance. Scores range from 0 to 12, with higher scores indicating better physical performance.
Fasting Blood Glucose | From enrollment to the end of treatment at 12 weeks.
  Measured to assess glycemic control before and after treatment.
2-Hour Postprandial Blood Glucose | From enrollment to the end of treatment at 12 weeks.
  Evaluated to further understand blood glucose management following meals.
Glycosylated Hemoglobin (HbA1c) | From enrollment to the end of treatment at 12 weeks.
  Measured to assess long-term glycemic control.
FRAIL Scale | From enrollment to the end of treatment at 12 weeks.
  Used to evaluate frailty status before and after the intervention, with scores indicating robustness, pre-frailty, or frailty.The FRAIL scale scores range from 0 to 5, with higher scores indicating greater frailty.
Rating of Perceived Exertion | Assessed after each training session, three times per week, throughout the 12-week treatment period.
  Assessed to gauge participants' subjective fatigue and exertion levels during training sessions.
Geriatric Depression Scale-15 | From enrollment to the end of treatment at 12 weeks.
  Measured to evaluate participants' psychological state and levels of depression before and after the intervention.The GDS-15 score ranges from 0 to 15, with higher scores indicating worse depressive symptoms.
Diabetes Distress Scale | From enrollment to the end of treatment at 12 weeks.
  Used to assess participants' distress related to diabetes management before and after treatment.Scores range from 1 to 6, with higher scores indicating greater distress related to diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- ZhejiangRongjun, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to share individual participant data (IPD) collected in this study, specifically including all relevant data sets that underpin the published results. This will encompass demographic information, clinical assessments, treatment responses, and outcome measures related to blood glucose levels, handgrip strength, gait speed, and psychological evaluations. The data will be de-identified to ensure participant confidentiality and will be made available to qualified researchers upon request after the study's completion. Sharing these data aims to promote transparency, facilitate further research, and enhance the understanding of the effects of Thera-Band elastic band-assisted progressive resistance-exercise training on patients with diabetes mellitus and frailty syndrome. Access will be subject to ethical review and data sharing agreements to protect participant privacy.
Supporting Information: Study Protocol
Time Frame: Individual participant data (IPD) and supporting information will be made available starting 6 months after the publication of the primary study results. This time frame allows for the completion of data analysis and publication processes. The data will remain accessible for a period of 5 years following the publication date to facilitate ongoing research and collaboration. During this time, interested researchers can request access to the IPD and any accompanying supporting information, subject to a data sharing agreement and ethical review to ensure participant confidentiality and proper use of the data.
Access Criteria: Access to individual participant data (IPD) and supporting information will be granted to qualified researchers and institutions for legitimate scientific research purposes, such as further analyses that build on the original study findings. Requests for access must be submitted in writing and will be reviewed by an independent Data Access Committee (DAC) comprised of study investigators and ethical experts. The DAC will evaluate requests based on criteria including the scientific merit of the proposed analysis, adherence to ethical standards, and feasibility of data sharing. Approved researchers will be required to sign a data sharing agreement that outlines the terms of use, including ensuring participant confidentiality and data protection measures. Access will be facilitated through a secure online platform where data can be accessed in compliance with relevant regulations and guidelines.

REFERENCES:
- [Derived] Ye M, Zhu Q, Yang H, Zhang L, Cai X. Effect of thera-band resistance training on diabetic patients with frailty syndrome. BMC Sports Sci Med Rehabil. 2025 Sep 29;17(1):284. doi: 10.1186/s13102-025-01350-9. PMID 41024136